CLINICAL TRIAL: NCT00369031
Title: A Phase I, Open Label, Parallel Group Trial To Evaluate Safety And Immunogenicity Of Three Nasal Immunisations Using A Fixed Dose-Level Of HIV gp140 V2 Loop Deleted Protein Adjuvanted With LTK63 Followed By Intramuscular Boosting With HIV gp140 V2 Loop Deleted Protein Adjuvanted With MF59 When Administered To Healthy Adults
Brief Title: Safety Study Of Nasal HIV Vaccine Adjuvanted With LTK63
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Safety issues
Sponsor: St George's, University of London (Other)
Collaborators: Richmond Pharmacology Limited (Industry); Novartis Vaccines (Industry); European Union (Other)
Responsible Party: David Lewis, Principal Investigator, SGUL
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2005-005983-10; C86P1; FP6-2002-LIFESCIHEA-2.3 503240
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Last update posted 2008-04-15 (Estimated); Status verified 2008-04

CONDITIONS: HIV Infections
Keywords: HIV; vaccine; nasal immunization
MeSH Terms: conditions — HIV Infections | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Human Immunodeficiency Virus glycoprotein 140 (vaccine)
  Interventions: Biological: Human Immunodeficiency Virus glycoprotein 140 (vaccine)
- 2 (Active Comparator): Human Immunodeficiency Virus glycoprotein 140 (vaccine) + Labile Toxin mutant LTK63 adjuvant
  Interventions: Biological: HIV glycoprotein 140 + Labile Toxin mutant LTK63 adjuvant
- 3 (Active Comparator): Labile Toxin mutant LTK63 adjuvant
  Interventions: Biological: Labile Toxin mutant LTK63 adjuvant

INTERVENTIONS:
Biological: Human Immunodeficiency Virus glycoprotein 140 (vaccine) — Human Immunodeficiency Virus glycoprotein 140 (vaccine) alone nasally
  Arms: 1
Biological: HIV glycoprotein 140 + Labile Toxin mutant LTK63 adjuvant — Human Immunodeficiency Virus glycoprotein 140 (vaccine) + Labile Toxin mutant LTK63 adjuvant nasally
  Arms: 2
Biological: Labile Toxin mutant LTK63 adjuvant — Labile Toxin mutant LTK63 adjuvant alone
  Arms: 3

SUMMARY:
The purpose of this study is to determine whether an HIV vaccine given as three nasal immunisations with a protein from HIV virus mixed with a toxoid adjuvant, followed by two intramuscular immunisations with the same protein mixed with a liquid adjuvant, causes untoward adverse reactions when administered to healthy adult volunteers. An initial evaluation of immune responses to the vaccine will also be undertaken.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether an HIV vaccine given as three nasal immunisations with a protein from HIV virus mixed with a toxoid adjuvant, followed by two intramuscular immunisations with the same protein mixed with a liquid adjuvant, causes untoward adverse reactions when administered to healthy adult volunteers. An initial evaluation of immune responses to the vaccine will also be undertaken by measuring gp140- and LTK63-specific IgG and IgA in cervical secretions, vaginal secretions, serum and nasal wash. IFNg secretion of T cells in response to gp140 peptide stimulation will be undertaken along with neutralising assays.

ELIGIBILITY:
Inclusion Criteria:

* They are adult volunteers, 18 to 45 years of age, who have signed an informed consent form following a detailed written explanation of participation in the protocol.
* They are volunteers who are in good health as determined by medical history, physical examination and clinical judgement.
* They are available for the duration of the study
* They are women who, if capable of becoming pregnant during the study, have agreed to have a pregnancy test immediately before immunisation, and to use appropriate contraception methods during the whole study period.

Exclusion Criteria:

* They have hypersensitivity to any component of the vaccines used in this study.
* They are found to be HIV antibody positive at the time of initial screening
* They have a known or suspected history of nasal disease, malignancy or abnormality, or any nasal disease, malignancy or abnormality discovered at time of screening.
* They have a known or suspected history of severe seasonal allergies and allergic rhinitis (requiring medication), recurrent nose bleeds, asthma, or cardio-pulmonary disease, or any of these conditions discovered at time of screening.
* They present in the samples obtained at the screening visit:
* a clinically significant amount of protein or haemoglobin in the urine sample, determined by urine dipstick:
* a clinically significant abnormality in the haematological or biochemical assays
* An abnormal value will be defined by the ranges quoted in the St George's Pathology Services Handbook.
* They have a known impairment of immune function or are receiving immunosuppressive therapy (including systemic or inhaled steroids, but excluding topical).
* They are receiving any medications via nasal route.
* They have any acute infections (including fever greater than or equal to 38°C) or any chronic disease.
* They are women capable of becoming pregnant who do not agree to have pregnancy testing before application of study products, or who do not agree to take appropriate contraception measures during the whole study period. Appropriate contraception shall include physician-prescribed oral, injected or implanted hormonal agents; barrier contraceptives used in conjunction with spermicidal agents; or intrauterine devices only.
* They present a current problem with substance abuse or with a history of substance abuse which, in the opinion of the investigator, might interfere with participation in the study.
* They have any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives.
* They have received an investigational agent within 3 months prior to study entry.
* They cannot speak fluent English, or are planning to leave the area of the study site prior to the end of the study period, or are likely not to complete the study.
* They have a weight (W)/height (H) index (WHI) less than 18.5 or greater than 40

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2006-09; Primary Completion 2007-11 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
To determine the frequency of vaccine-related local and systemic adverse events after nasal immunisation up to week 32 | 32 weeks

SECONDARY OUTCOMES:
To determine the frequency of vaccine-related local and systemic adverse events after intramuscular immunization up to week 32 | 32 weeks
To determine the frequency of subjects mounting a serum IgG neutralising antibody response to gp140 at weeks 0, 4, 8, 10, 12, 16, 28 & 32 | 32 weeks
To determine the frequency of subjects mounting a nasal wash gp140-specific IgA response to gp140 at weeks 0, 4, 8, 10, 12, 16, 28 & 32 | 32 weeks
To determine the frequency of female subjects mounting a vaginal secretions IgA response to gp140 at weeks 0, 4, 8, 10, 12, 16, 28 & 32 | 32 weeks
To determine the frequency of subjects with a serum T-cell response to gp140 at weeks 0, 4, 8, 10, 12, 16, 28 & 32 | 32 weeks
To determine frequency of subjects mounting a serum IgG response, nasal IgA response and vaginal IgA response to LTK63 at weeks 0, 4, 8, 10, 12, 16, 28 & 32 | 32 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David JM Lewis, MD, Principal Investigator — St George's, University of London, UK
Locations (1):
- St George's Vaccine Institute, London, England, United Kingdom

REFERENCES:
- See also: St George's Vaccine Institute Home website — http://www.vaccine.ac.uk